CLINICAL TRIAL: NCT02206230
Title: A Randomized Controlled Trial of Conventional Versus Hypofractionated Radiation Therapy With Temozolomide for Patients With Newly Diagnosed Glioblastoma
Brief Title: Trial of Hypofractionated Radiation Therapy for Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR-02-1401
Record Dates: First submitted 2014-07-24; First posted 2014-08-01 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Glioblastoma
Keywords: glioblastoma; radiotherapy; hypofractionated radiotherapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: 1:1, randomized, open label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypofractionated radiation therapy (Experimental): Hypofractionated radiation therapy of 60 Gy in 20 fractions (3 Gy per fraction) with concurrent temozolomide 75 mg/m2 given 7 days/week. After a 4-week break, temozolomide days 1-5 every 28 days for 6-12 cycles(as per institutional standard)..
  Interventions: Radiation: Hypofractionated radiation therapy
- Standard radiation therapy (Active Comparator): Standard radiation therapy of 60 Gy in 30 fractions (2 Gy per fraction) with concurrent temozolomide 75 mg/m2 given 7 days/week. After a 4-week break, temozolomide days 1-5 every 28 days for 6-12 cycles(as per institutional standard)..
  Interventions: Radiation: Standard radiation therapy

INTERVENTIONS:
Radiation: Hypofractionated radiation therapy
  Arms: Hypofractionated radiation therapy
Radiation: Standard radiation therapy
  Arms: Standard radiation therapy

SUMMARY:
This study is being done to compare standard radiation therapy with hypofractionated radiation therapy for patients with newly diagnosed glioblastoma

DETAILED DESCRIPTION:
Hypofractionated radiation therapy (RT) in the treatment of patients with glioblastoma, 18 - 70 years of age with good performance status (ECOG 0 - 2), will be well tolerated and yield survival non-inferior to conventional fractioned RT, allowing significant abbreviation of the length of the radiation course required for these patients with limited survival. The importance of hypofractionation is, therefore, not in improving survival, but rather to shorten RT duration to improve patient comfort and convenience. This approach is pertinent given the limited life expectancy of glioblastoma and has been used in patients with prolonged survival including breast and prostate cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Newly-diagnosed, histologically proven, intracranial glioblastoma or gliosarcoma treated with maximal safe resection, which may be biopsy alone if resection is not possible.
2. History and physical examination, including neurological examination, within 14 days prior to randomization.
3. Age between 18 and 70 years, inclusive.
4. ECOG performance score 0-2.
5. Stable or decreasing dose of corticosteroids for at least 14 days prior to randomization (Stupp et al.).
6. Laboratory evaluation obtained within 7 days prior to randomization, with adequate function as defined below: (Stupp et al.)

   1. ANC ≥ 1.5 x 10^9/L
   2. Platelets ≥ 100 x 10^9/L
   3. Serum creatinine ≤ 1.5 times ULN
   4. Total serum bilirubin ≤ 1.5 times ULN
   5. ALT < 3 times ULN
   6. AST < 3 times ULN
   7. Alkaline phosphatase < 3 times ULN
7. Patients must sign a study-specific informed consent prior to study registration and must be willing to comply with study treatment, questionnaire completion and follow-up.

Exclusion Criteria:

1. Recurrent or multifocal malignant gliomas. Multicentric gliomas, defined as multiple, discrete areas of enhancement on T1 weighted MRI sequences with contrast all contained within one connected region of abnormality on T2 weighted/FLAIR MRI sequences, are allowed to enroll on this study.
2. Prior invasive malignancy (except for non-melanomatous skin cancer) unless expected survival from prior malignancy is ≥ 5 years.
3. Prior head or neck RT (except for T1 glottic cancer), or systemic therapy precluding delivery of concurrent and adjuvant temozolomide
4. Treatment with any other therapeutic clinical protocol within 30 days prior to study registration or during participation in the study.
5. Severe, active co-morbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization
   2. Transmural myocardial infarction within the last 6 months
   3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study registration
   4. Any severe, active co-morbidity precluding delivery of temozolomide.
6. Women of child-bearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
7. Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant due to temozolomide.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-09-25 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Overall survival | Patients without an event will be censored the last time they were known to be alive. Median, 6-month, 1-year, and 2-year OS rates will be measured.
  defined as the time between randomization and death due to any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Patients without an event will be censored at date of last follow-up for progression. Patients with no post-baseline follow-up for progression will be censored at day of randomization. Median, 6-month, 1-yr, and 2-yr PFS rates will be measured
  defined as the time between randomization and radiographic progression based on RECIST criteria (see section 4.5) or clinical progression leading to institution or change in radiation or systemic therapy for progressive or recurrent disease or death due to any cause.
Adverse events according to NCI CTCAE version 4.0 criteria. | Evaluated weekly during radiation therapy; on C1D1 and at the end of every 2 cycles of adjuvant temozolomide; post-treatment follow-up every 4 months for 2 years, then every 6 months for years 3-5 up until progression/palliative
  Adverse events will be reported as listings and summarized as frequency tables. Additional reports by grade, causality, and relationship to study treatment will be produced. Incidence of adverse events by stratification variables will be assessed
Health-related quality-of-life as assessed by MMSE and EORTC QLQ-C30/QLQ-BN20 questionnaires. | Evaluated at baseline, weekly during radiation therapy, at the end of every 2 cycles of adjuvant temozolomide, and post-treatment follow-up every 4 months for 2 years, then every 6 months for years 3-5 up until progression/palliative
  Kaplan-Meier curves and estimates of median time to event, and corresponding 95% confidence intervals, for each health-related quality-of-life scale (overall score of MMSE and each measure on EORTC QLQ-C30/QLQ-BN20 questionnaires) will be assessed. The difference in health-related quality-of-life between the treatment arms will be determined with a stratified log-rank test at the 5% alpha level

CONTACTS AND LOCATIONS:
Overall Officials: Samir Patel, MD, Principal Investigator — Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Yang F, Dinakaran D, Heikal AA, Yaghoobpour Tari S, Ghosh S, Amanie J, Murtha A, Rowe LS, Roa WH, Patel S. Dosimetric predictors of toxicity in a randomized study of short-course vs conventional radiotherapy for glioblastoma. Radiother Oncol. 2022 Dec;177:152-157. doi: 10.1016/j.radonc.2022.10.016. Epub 2022 Oct 20. PMID 36273738